CLINICAL TRIAL: NCT02934490
Title: The Effect of New-style Vaginal Repair Mesh in the Treatment of Female Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinan Military General Hospital (Other)
Responsible Party: Principal Investigator, Geping Yin, Director, Jinan Military General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013ZX05
Record Dates: First submitted 2016-09-23; First posted 2016-10-17 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Surgical Mesh

ARMS (1):
- Treatment group (Experimental)
  Interventions: Device: Mesh

INTERVENTIONS:
Device: Mesh — Meshes were made by Gynemech TM PS, (Johnson & Johnson Shanghai Medical Equipment Co. SFDA registration No. 3460365, size 10 × 15cm)

SUMMARY:
The study is to explore the effectiveness of a new-style anterior vaginal wall mesh in the treatment of female stress urinary incontinence(SUI). Meshes were made by Gynemech TM PS, (Johnson & Johnson Shanghai Medical Equipment Co. China Food and Drug Administration (CFDA) registration No. 3460365, size 10 × 15cm). Meshes were cut to appropriate size. The incontinence questionnaire summary table (ICIQ-SF), pad test, urodynamic and other diagnostic tests were used for preoperative assessment and the evaluation of postoperative surgical outcome and complication. The results were compared with the one-year cure rates of Burch and trans vaginal taping (TVT) surgeries. The analysis indicated that the surgery using the new-style anterior vaginal mesh, as a minimally invasive procedure, not only achieved its expectation with similar cure rate to Burch, TVT/ trans vaginal taping obturator (TVT-O) surgeries, but also has lower economic cost and complication rate than the TVT /TVT-O approach. The evaluation of long-term treatment effect needs further follow-up of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically and biopsy confirmed non-neoplastic lesions of genital skin and mucous membrane (non-neoplasia epithelial disorders of skin and mucosa of vulva). Symptoms include repeated itching, discoloration, rhagades, loss of skin elasticity and dyspareunia that affect the patients' quality of life.

Exclusion Criteria:

* Atypical hyperplasia or vulvar cancer confirmed by biopsy of genital lesions;
* Vulvovaginal or other gynecological trauma, acute inflammatory diseases and other acute illness in need of urgent care;
* Combined with other serious gynecological diseases (symptomatic hysteromyoma, ovarian tumor, etc.), and/or severe organ diseases (such as heart, lung, brain and renal disease/failure) that need immediate treatment;
* Other type of cancers that require urgent care.

Ages: 27 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2009-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Anatomy of female perineal bilateral pubic bones | Two months before treatment
  Anatomy of the main parameters of bilateral gap: female perineum pubis bilateral acupoint location, angle, length and width of the acupuncture points.
Anatomy of female perineal bilateral pubic bones | One month after treatment
  Anatomy of the main parameters of bilateral gap: female perineum pubis bilateral acupoint location, angle, length and width of the acupuncture points.
Incontinence questionnaire summary table observation | Three months before treatment
  Incontinence questionnaire summary observation to evaluate the therapeutic effect of the study on the implantation of mesh in female stress urinary incontinence. If there are complications, including the cough so, sneezing or laughing, and lifting whether there is leakage of urine and preoperative contrast, whether the situation is better; whether the quality of life. The increase; whether the foreign body discomfort; and other discomfort.
Incontinence questionnaire summary table observation | Six months after treatment
  Incontinence questionnaire summary observation to evaluate the therapeutic effect of the study on the implantation of mesh in female stress urinary incontinence. If there are complications, including the cough so, sneezing or laughing, and lifting whether there is leakage of urine and preoperative contrast, whether the situation is better; whether the quality of life. The increase; whether the foreign body discomfort; and other discomfort.
Incontinence pad weight test | Three months before treatment
Incontinence pad weight test | Six months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Military General Hospital, Jinan, Shandong, China

REFERENCES:
- [Derived] Yin G, Yuan Z, Li J, Liang J, Wu A, Liu N. A new treatment of female stress urinary incontinence with vaginal antetheca-retropubic space mesh repair surgery: a clinical trial. World J Urol. 2018 Jul;36(7):1103-1109. doi: 10.1007/s00345-018-2234-6. Epub 2018 Feb 24. PMID 29478148